CLINICAL TRIAL: NCT05285228
Title: Motivational Effect of Choosing the Taste of te Fluoride Varnish on Acceptance and Behavior During Dental Visit in Children - a Single Blind RCT
Brief Title: Motivational Effect of Choosing Taste of te Fluoride Varnish on Behavior During Dental Visit in Children - RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BB 180/21
Record Dates: First submitted 2022-02-15; First posted 2022-03-17 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Child Behavior
Keywords: cooperation; pediatric dentistry; behavior management; fluoride varnish
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor enters the room to observe the dental treatment after the allocation to the group when the fluoride varnish is placed ready.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: allocation to specific taste of fluoride varnish (Active Comparator): allocation to specific taste of fluoride varnish
  Interventions: Behavioral: given fluoride varnish (control)
- Test group: child chooses taste of fluoride varnish (Experimental): child chooses taste of fluoride varnish before dental treatment
  Interventions: Behavioral: effect of choice on cooperation (pseudoalternative)

INTERVENTIONS:
Behavioral: effect of choice on cooperation (pseudoalternative) — For the test group, before the standard check-up starts, the participant is given the choice of selecting the taste of the fluoride varnish (Profluorid VOCO, Germany) from a range of about five flavors (Melon, Caramel, Cherry, Bubble gum, Mint), which will be applied at the end of the visit. Post-placement instructions provided by the manufacturer will be given to the caregiver and the child and questionnaires will be handed out.
  Other Names: fake alternative
  Arms: Test group: child chooses taste of fluoride varnish
Behavioral: given fluoride varnish (control) — For the control group the participant is provided with a given taste of the fluoride varnish (Profluorid VOCO, Germany) from a range of about five flavors (Melon, Caramel, Cherry, Bubble gum, Mint) according to the randomization list.
  Arms: Control group: allocation to specific taste of fluoride varnish

SUMMARY:
To assess the influence of the choice of fluoride varnish flavor on the acceptance and cooperation in schoolchildren between (5-10) years during the dental visit, in which an application of fluoride varnish is indicated.

DETAILED DESCRIPTION:
The main assumption of the study is giving the child the option to choose e.g. their preferred taste of the fluoride varnish possibly moves the focus away from not being willing to receive the fluoride varnish application to rather accepting it (pseudoalternative).

The aim of this study is to investigate the impact of participation via choosing the taste of the fluoride varnish (locus of control and pseudo-alternative) on the acceptance and cooperation during dental visit in schoolchildren aged 5 to 10 years.

This two-parallel arm single-blind randomized controlled clinical trial will be undertaken at the Department of Preventive and Pediatric Dentistry at the University of Greifswald from approximately January 2022 to Autumn 2022. The child will be randomly allocated using simple random sampling with the use of random table method, in which 35 randomly generated serial numbers for each group will be generated by Windows Microsoft Excel (2010, USA) to ensure equal randomization of each group.

The test group will receive a previously allocated flavor of fluoride varnish (Profluorid VOCO, Germany) ranging from (Melon, Caramel, Cherry, Bubble gum, Mint) containing 22,500 ppm fluoride. However the test group will be receiving the choosing the taste of the previously mentioned fluoride varnish r with flavor ranging from (Melon, Caramel, Cherry, Bubble gum, Mint). After allocation an independent observer enters the dental treatment room for blinded assessment. After the dental visit, the participating child, the accompanying parent or caregiver, the dental operator and the blinded assessor receive a short questionnaire to be filled out.

Patients presenting with acute pain or with signs and symptoms, which should be treated will not be asked to participate. Moreover Systemic diseases that require special attention during their dental treatment or Parents/children who refused to participate in the study, and reported allergy against ingredients of the toothpaste are excluded from participation.

Assessment would be done firstly by observing participants' behavior and then categorized using the Frankl's behavior rating scale-FRS (Frankl, 1962) by an independent blinded observer, and the accompanying parent.

Secondly, The dental anxiety level of the child using the facial image scale (FIS) consists of a row of five gray scale faces ranging from very happy to very unhappy, moreover a questionnaire will be filled out by the caregivers (including questions on demographic issues) on their acceptance and preference regarding the choice of the taste of the fluoride varnish.

Further data of the child for better description of the baseline characteristics of the participants will be taken from the documentation in the patient's file: e.g. age, sex, dmft / DMFT, history of dental anxiety, history of invasive dental treatment e.g. nitrous oxide sedation or dental general anesthesia.

ELIGIBILITY:
Inclusion criteria

* Children aged between 5 - 10 years.
* Clinical presentation due to a dental appointment, in which an application of fluoride varnish is planned.

Exclusion criteria

* Patients presented with acute pain/ patients with signs or symptoms to be treated.
* Patients reported with systemic diseases that require special attention during their dental treatment.
* Parents or children, who refuse participation in the study.
* Reported Allergy against ingredients of the toothpaste or the fluoride varnish.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
acceptance of dental treatment | assessment during the dental visit via independent observer; usually the dental visit does not exceed more than 30 minutes; the overall behavior is rated during this time period
  measurement via Frankl behavioral scale;

SECONDARY OUTCOMES:
acceptance of taste of fluoride varnish | assessment right after the end dental visit by the child; immediately, this means within about 1 minute after the application of the varnish
  patient rates the acceptance of the taste of the fluoride varnish with a facial image scale (from definitely negative to definitely positive: codes 1 to 5)

OTHER OUTCOMES:
parental acceptance regarding the use of the fluoride varnish | questionnaire is filled out right after the end of the dental visit by the parent, immediately, this means within about 1 minute after the application of the varnish
  parents receive a simple questionnaire with 10 items and a rating scale (from 1-5 each). 4 sociodemographic characteristic aspects are included as gender, age and level of education

CONTACTS AND LOCATIONS:
Overall Officials: Karim Ramiar, Principal Investigator — University of Greifswald
Locations (1):
- Dental Clinics University of Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karim R, Splieth CH, Schmoeckel J. Effect of Choice of Flavor of Fluoride Varnish on Behavior in Dental Visits in Schoolchildren. Clin Exp Dent Res. 2025 Feb;11(1):e70069. doi: 10.1002/cre2.70069. PMID 39898776